CLINICAL TRIAL: NCT05529238
Title: Effectiveness of Supervised Kegel Exercises Using Bio-feedback Versus Unsupervised Kegel Exercises on Stress Urinary Incontinence: A Quasi-experimental Study
Brief Title: Kegel Exercises for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Darwin University (Other)
Responsible Party: Principal Investigator, Donelle Cross, Lecturer, Charles Darwin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interventional
Record Dates: First submitted 2022-08-26; First posted 2022-09-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supervised group during study (Other): monthly physiotherapist appointment for half of the cohort including pelvic floor examination by physiotherapist including digital palpation and perineometry.
  Interventions: Behavioral: biofeedback training
- unsupervised group during study (No Intervention): No intervention. Participants to practice kegel exercises at home.

INTERVENTIONS:
Behavioral: biofeedback training — participants received biofeedback training for kegel exercises in the supervised group. the unsupervised group practised their Kegel exercises at home
  Arms: supervised group during study

SUMMARY:
Study about a targeted group of women suffering from self-reported stress urinary incontinence, attend a Kegel exercise training program. The group was divided into two; supervised and unsupervised. Whilst both groups benefited from initially seeing a women's health physiotherapist for a pelvic floor muscle assessment and a bespoke Kegel exercise program, only the supervised group continued to see the physiotherapist for monthly bio-feedback training. The unsupervised group relied on their own motivation to perform their Kegel exercises as prescribed. At the end of the twelve week program, both groups had a final pelvic floor muscle strength assessment by the physiotherapist to determine any changes and subsequent improvements in urinary incontinence.

Aim : Investigate and compare the efficacy of supervised Kegel exercises with biofeedback on Stress Urinary Incontinence (SUI) and Pelvic Floor Muscle Strength (PFMS) compared to unsupervised Kegel exercises.

The primary goal of this study was to determine the effectiveness of supervised Kegel exercises using BT versus unsupervised Kegel exercises without biofeedback training, on SUI. A secondary outcome was to establish whether an improvement was observed in PFMS and subsequently, the effect of this on SUI. It was hypothesized that regular support and visual motivation and direction of BT from the physiotherapist, would provide greater results.

ELIGIBILITY:
Inclusion Criteria:

* being female
* aged over 18 years
* suffer from SUI (their subjective disclosure was based on a description provided for their reference)
* did not perform Kegel exercises
* be available for duration of 12-week program

Exclusion Criteria:

* pregnancy and breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — must be female
Enrollment: 29 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-08-18 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Incontinence severity index (ISI) tool | Week 0
  self-reported questionnaire describing frequency/severity of urinary incontinence. the higher the number, the higher the impact.
Incontinence severity (ISI) index tool | Week 12
  self-reported questionnaire describing frequency/severity of urinary incontinence. the higher the number, the higher the impact.
Pelvic floor assessment from physiotherapist | week 0
  pelvic floor muscle strength
Pelvic floor assessment from physiotherapist | week 12
  pelvic floor muscle strength

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Darwin University, Darwin, Northern Territory, Australia